CLINICAL TRIAL: NCT02310685
Title: The Canadian Health Improvement Network to Upgrade Prevention Services (CHIN-UPS) - Evaluating a Multidisciplinary Health Promotion Program.
Brief Title: the Canadian Health Improvement Network to Upgrade Prevention Services
Acronym: CHIN-UPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Steven Grover, MD, Steven A. Grover, MD, MPA, FRCPC, McGill University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: A10-M75-14B
Record Dates: First submitted 2014-11-24; First posted 2014-12-08 (Estimated); Last update posted 2019-08-13 (Actual); Status verified 2019-08

CONDITIONS: Cardiovascular Disease
Keywords: Cardivascular risks (hypertension, sedentary, overweight); Cardiovascular age; E-health wellness program; Prevention; Community pharmacists; Lifestyle change; Cardiometabolic age
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension; Sedentary Behavior; Overweight

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Active Comparator: Intervention The primary focus is CVD risk factors. Subjects will be shown how to update Cardiovascular Age or Cardiometabolic Age on website. Pharmacists will give overview of comprehensive ehealth wellness program. Subjects will complete additional health assessments which include questionnaires considered gold standard. Pharmacists will explain that participants have access to ehealth coaching based educational modules with information relevant to a better understanding of cardiovascular risk factors. The ehealth coaching modules are guides to help understand risk factors and importance of making lifestyle changes. As information alone is often insufficient to promote change, participants will have access to online physical activity challenges.
  Interventions: Other: Comprehensive e-health wellness program
- No Intervention (No Intervention): Individuals randomized to the non active intervention group will have access to modified version of ehealth website. The pharmacist will show participants how to update Cardiovascular Age or Cardiometabolic Age on website. They will have access to health assessments but not ehealth coaching educational modules or challenges. They will have online support tools including public domain education material on exercise, healthy eating, understanding and managing blood pressure, diabetes and smoking cessation. Participants will return to the pharmacist for follow-up visits at 3, 6 months and one year. The pharmacist will update their cardiovascular risk profile with current information At the first follow up visit and at 1 year participants will be asked to have blood lipids reassessed.

INTERVENTIONS:
Other: Comprehensive e-health wellness program — Participants randomized to this arm will have complete access to the myhealthcheckup website equipped with online tools including health assessments with coaching modules, educational material with quizzes, exercise challenges and motivational tips. The subject will meet with the pharmacist on 4 occasions (initial, 3, 6, 12 months) to update the cardiovascular risk profile, BP, weight, waist circumference and lipid profile. All interventions that were prespecified to be administered as part of the protocol, even if a particular intervention is not "of interest".
  Arms: Intervention

SUMMARY:
RATIONALE Controlling cardiovascular risk factors has been proven to be effective in prevention and management of cardiovascular disease (CVD). Nonetheless, significant treatment gaps have been demonstrated repeatedly in numerous surveys. A recent study of Canadian adults filling prescriptions for hypertension or dyslipidemia demonstrated that the majority remained overweight and sedentary despite being at risk of developing CVD. Medication adherence has been shown to be poor with up to 50% of patients stopping therapy after one year.

Patient-centred care can lead to improved clinical management and patient satisfaction. Adherence with prescribed therapy can also be improved if individuals understand the importance of their risk factors, are aware of their overall health status and participate in decision making surrounding pharmacotherapy and lifestyle changes.

Community pharmacists are frontline healthcare professionals who can identify patients at risk of CVD, assess their adherence with recommended lifestyle behaviours or drug therapy and engage them in shared decision making surrounding health promotion strategies. Local pharmacies could effectively become readily accessible community health centres nationwide.

Research Objectives. The primary objective is to evaluate, in a randomized clinical trial, the impact of a community pharmacy intervention to improve the management of cardiovascular risk factors vs a basic e-health education program. The intervention will include a cardiovascular or cardiometabolic risk assessment providing the individual with their Cardiovascular or Cardiometabolic Age. Individuals at increased risk of CVD and/or with modifiable risk factors will also be offered a one year subscription to a multidisciplinary, pharmacy based, e-health promotion program to improve management of CVD risk factors such as weight loss and increased physical activity and track their progress in managing their risk factors and reducing their Cardiovascular or cardiometabolic Age. Changes in CVD risk factors, Cardiovascular/cardiometabolic Age, and uptake or adherence to medications and lifestyle changes will be examined 3 months, 6 months and one year post intervention.

Study Hypothesis. Investigators hypothesize that engaging patients in a discussion of their Cardiovascular or Cardiometabolic Age and management of their risk factors will result in improved healthy lifestyle habits moreover increased physical activity and weight loss.

DETAILED DESCRIPTION:
Twelve hundred subjects will be recruited from 30 to 60 pharmacies across Canada each providing 20 to 40 study subjects. Recruitment will occur over 18 months.

Shoppers Drug Mart and Sobeys/Lawtons are chain pharmacies that have agreed to participate in the study and will identify a minimum of 20 and 10 pharmacies from within their chains respectively. Pharmacy contacts will be sent summary of the research project and will be invited to participate by senior management through internal company communications. Additional pharmacies will be included in the study if additional funding to remunerate the pharmacists becomes available.

A pharmacy will be eligible to participate if it has an automated blood pressure system, a calibrated weight scale, a consultation area with a computer, internet access and the pharmacist is willing to recruit and enroll at least 20 patients.

Once a pharmacist has agreed to participate, pharmacist will be asked to participate in a conference call. A one-hour training webinar will be provided to the pharmacists prior to initiating recruitment. Each pharmacist will have access to the website so that pharmacist can try the health assessments, read the e-health coaching educational modules and personally participate in the health challenges. Pharmacist will be given access to a series of online training modules for cardiovascular/cardiometabolic risk assessments and how to engage patients to improve lifestyle behaviours such as exercise, weight loss and smoking cessation. Pharmacists responsibilities will include taking the participant's blood pressure, weight and waist measurements and enabling the participant to get recent blood lipids. The pharmacist will also interpret their cardiovascular/cardiometabolic risk profile and provide patient with the appropriate educational materials. This visit is expected to take 20-25 minutes. Pharmacists will also be encouraged to have participants return for follow-up visits every 3 months to discuss strategies to achieve their behaviour change goals and review results.

Subjects will be recruited by the pharmacist or pharmacy staff using number of strategies.

1. Study recruitment will be promoted within each pharmacy using flyers and posters. Any individual at increased cardiovascular risk who is interested in reducing their cardiovascular risk by losing excess body weight or increasing their fitness level will be encouraged to view study information and register directly on the website.
2. Individuals who are sedentary, overweight will be invited to enroll in the study by registering on website.
3. Recruited subjects can promote the program to friends and family members. In such cases, they will be allocated to the same treatment group.

Study procedures Individuals will be invited to register on myhealthcheckup website. Access to their account will be limited to the participant, members of the research team and their local pharmacist. Those who are interested in participating will be asked to sign the online informed consent form. Participants will be asked to complete a health assessment for heart/diabetes and fitness. Included in this assessment are two validated questionnaires including The International Physical Activity Questionnaire and the Self-Efficacy for Lifestyle Behaviour Change Questionnaire and the questions required to determine if the participant can exercise safely. Additional health assessments will be completed at study entry and all of the assessments will be repeated at 3 months, 6 months, and one year post intervention.

Once the individuals have registered, signed Informed Consent Form and completed the myhealthcheckup assessments, participants will select their pharmacist from a list provided on the website and they will schedule their initial appointment with their pharmacist. Selecting a health coach or pharmacist is optional.

The initial visit with the pharmacist will take approximately 20 to 25 minutes. During this visit, participants will be informed that more than one intervention is being evaluated and that they have been randomly assigned to only one. More specifically, they have been assigned to either the comprehensive e-health wellness program or the basic e-health education program. Randomization will occur at registration. The pharmacist will take the patient's blood pressure, weight and waist measurements, will interpret the patient's cardiovascular/cardiometabolic risk profile and discuss a plan of action. Each participant will be provided with baseline cardiovascular or cardiometabolic risk assessment. Both the active intervention and the non-active intervention groups will have access to their cardiovascular or cardiometabolic risk profile, including their calculated cardiovascular/cardiometabolic age. It provides their estimated 10-year risk of developing cardiovascular disease and compares this result to Canadians of the same age and gender. The risk profile will be interpreted by pharmacist.

Most of the information required for baseline cardiovascular risk assessment will be provided by the participant. Clinical information will include: age, gender, presence of previously diagnosed cardiovascular diseases including coronary heart disease, cerebrovascular disease or lower extremity peripheral arterial disease; previously diagnosed diabetes, family history of premature cardiovascular disease, smoking status, use of antihypertensive medication and self-reported weekly exercise. Required clinical information includes resting blood pressure, height, weight, waist circumference, and non-fasting cholesterol values. Blood pressure will be measured. When actual lipid values are not known, the Framingham and Cardiovascular Age risk profiles will be completed using the median lipid values for Canadians of same age and gender and each participant will be told to ask their doctor for most recent values to update their record and allow a more accurate risk assessment to be completed by the patient at home online (intervention group only) or during their next visit to the pharmacy. This initial visit should take 20-25 minutes.

Both groups of patients will be asked to return to their pharmacist after 3 months, 6 months and 1 year for follow-up visit to have their cardiovascular risk profile updated. At each visit, blood pressure, weight and waist circumference will be measured and any changes in other risk factors will be noted. Each participant's progress will be evaluated during the follow-up visits.

Active Intervention: Comprehensive e-health wellness program Given the primary focus on CVD risk factors, each subject will be shown by the pharmacist how to update their Cardiovascular or Cardiometabolic Age on website. Pharmacists will give subjects brief overview of what the comprehensive e-health wellness program website has to offer them. Patients will be shown that in addition to the cardiovascular or cardiometabolic risk, diabetes and fitness assessments, they will be able to complete eight additional health assessments at entry into the study and as they see fit. All of the assessments employ questionnaires considered the gold standard for evaluating each of the respective health conditions which include: 1) smoking and nicotine dependence 2) alcohol abuse and dependence 3) sleep 4) depression 5) stress 6) fitness 7) nutrition and 8) body weight. Subjects will have access to summary of health status results and identify where there is room for improvement according to current disease treatment guidelines.

The pharmacist will explain that participants have access to ehealth coaching based educational modules with information relevant to a better understanding of exercise, weight loss, hypertension, dyslipidemia and diabetes and how to improve other areas such as sleep, stress management, and smoking cessation. The goal of these ehealth coaching modules are designed to encourage the individual to remain engaged and to take charge of their physical and mental health by increasing their physical activity, making healthy food choices and learning tools to decrease stress and improve sleep habits. Participants will receive daily health tips.

As information alone is often insufficient to promote behaviour change, participants will have access to online physical activity challenges designed to motivate the user to engage in regular exercise. The challenges provide tracking tools to facilitate the subject's monitoring of their progress. Physical activity challenges can be designed to engage the subject as a member of an online team. Participants can also compete individually in specific challenges. Individuals participating in a team challenge will be asked to provide a pseudonym to protect anonymity. Participants will have 24/7 access to their health record and be encouraged to use the website to evaluate a range of health assessments, receive information about specific health conditions, or engage in the online activity challenges. Subjects can review what the pharmacist explained to them concerning the website by viewing a brief video that will be provided on the website home page.

Non-active intervention: Basic e-health education program Individuals randomized to the non-active intervention group will be provided with access to a modified version of the e-health website.

Each participant will be shown by the pharmacist how to update their Cardiovascular Age or Cardiometabolic Age on the website. Participants will have access to other health assessments but not the ehealth coaching based educational modules or the challenges. Instead participants will be provided on-line support tools including public domain education material such as handouts on exercise, healthy eating, understanding and managing blood pressure, diabetes and smoking cessation. These are currently available from the Public Health Association of Canada. Participants will be asked to see their pharmacist for a follow-up visit at 3 months, 6 months and one year. During these visits the pharmacist will update participants' cardiovascular or cardiometabolic risk profile with current clinical information including a measured blood pressure and weight. At the first follow-up visit and at 1 year, all participants will be asked to have their blood lipids re-assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 40-75 years
2. Overweight defined as BMI > 27
3. Sedentary Lifestyle (less than 3 hours of moderate physical activity per week)
4. Access to Internet daily
5. Speak and read English or French

Exclusion Criteria:

1. Unable to sign informed consent
2. Pregnant
3. Have a health condition that would exclude them from being able to safely lose 10 lbs if their BMI is >27 kg/m2 OR to exercise daily at a moderate intensity (equivalent to brisk walking) for at least 30 minutes

Note: All individuals are eligible to participate in the program; however only those who meet the inclusion criteria will be included in the analysis. Those who meet the exclusion criteria will not be included in the analysis. Pregnant women and individuals who answered yes to the safety questionnaire will receive the following message on the website and in an email: If you answered yes to any of the exercise safety questions, we recommend that you obtain clearance from your physician prior to changing your exercise program. Individuals will tick a box "I have read this message"

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 459 (Actual)
Dates: Start 2015-01; Primary Completion 2018-09 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Weight loss/exercise | April 2015 to October 2017, up to 28 months
  Weight loss/exercise will be measured and assessed at 3, 6, and 12 months.

SECONDARY OUTCOMES:
Blood Pressure | April 2015 to October 2017, up to 28 months
  Blood pressure will be measured at baseline, 3, 6 and 12 months.
Drop-out rates | April 2015 to October 2017, up to 28 months
  drop out rates in each arm
Medication adherence | April 2015 to October 2017, up to 28 months
  Medication adherence will be analysed

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Grover, MD MPA FRCPC, Principal Investigator — McGill University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grover SA, Lowensteyn I, Joseph L, Kaouache M, Marchand S, Coupal L, Boudreau G. Discussing coronary risk with patients to improve blood pressure treatment: secondary results from the CHECK-UP study. J Gen Intern Med. 2009 Jan;24(1):33-9. doi: 10.1007/s11606-008-0825-4. Epub 2008 Oct 21. PMID 18937013
- [Background] Heatherton TF, Kozlowski LT, Frecker RC, Fagerstrom KO. The Fagerstrom Test for Nicotine Dependence: a revision of the Fagerstrom Tolerance Questionnaire. Br J Addict. 1991 Sep;86(9):1119-27. doi: 10.1111/j.1360-0443.1991.tb01879.x. PMID 1932883
- [Background] Saunders JB, Aasland OG, Babor TF, de la Fuente JR, Grant M. Development of the Alcohol Use Disorders Identification Test (AUDIT): WHO Collaborative Project on Early Detection of Persons with Harmful Alcohol Consumption--II. Addiction. 1993 Jun;88(6):791-804. doi: 10.1111/j.1360-0443.1993.tb02093.x. PMID 8329970
- [Background] Bastien CH, Vallieres A, Morin CM. Validation of the Insomnia Severity Index as an outcome measure for insomnia research. Sleep Med. 2001 Jul;2(4):297-307. doi: 10.1016/s1389-9457(00)00065-4. PMID 11438246
- [Background] Myers JK, Weissman MM. Use of a self-report symptom scale to detect depression in a community sample. Am J Psychiatry. 1980 Sep;137(9):1081-4. doi: 10.1176/ajp.137.9.1081. PMID 7425160
- [Background] Cohen S, Kamarck T, Mermelstein R. A global measure of perceived stress. J Health Soc Behav. 1983 Dec;24(4):385-96. No abstract available. PMID 6668417
- [Background] Craig CL, Marshall AL, Sjostrom M, Bauman AE, Booth ML, Ainsworth BE, Pratt M, Ekelund U, Yngve A, Sallis JF, Oja P. International physical activity questionnaire: 12-country reliability and validity. Med Sci Sports Exerc. 2003 Aug;35(8):1381-95. doi: 10.1249/01.MSS.0000078924.61453.FB. PMID 12900694
- [Background] Gans KM, Risica PM, Wylie-Rosett J, Ross EM, Strolla LO, McMurray J, Eaton CB. Development and evaluation of the nutrition component of the Rapid Eating and Activity Assessment for Patients (REAP): a new tool for primary care providers. J Nutr Educ Behav. 2006 Sep-Oct;38(5):286-92. doi: 10.1016/j.jneb.2005.12.002. PMID 16966049
- [Result] Grover S, Coupal L, Kouache M, Lowensteyn I, Marchand S, Campbell N. Estimating the benefits of patient and physician adherence to cardiovascular prevention guidelines: the MyHealthCheckup Survey. Can J Cardiol. 2011 Mar-Apr;27(2):159-66. doi: 10.1016/j.cjca.2011.01.007. PMID 21459263
- [Result] Grover SA, Lowensteyn I, Joseph L, Kaouache M, Marchand S, Coupal L, Boudreau G; Cardiovascular Health Evaluation to Improve Compliance and Knowledge Among Uninformed Patients (CHECK-UP) Study Group. Patient knowledge of coronary risk profile improves the effectiveness of dyslipidemia therapy: the CHECK-UP study: a randomized controlled trial. Arch Intern Med. 2007 Nov 26;167(21):2296-303. doi: 10.1001/archinte.167.21.2296. PMID 18039987
- See also: myhealthcheckup website — https://www.google.ca/#q=myhealthcheckup